CLINICAL TRIAL: NCT05357690
Title: Stellate Ganglion Blockade for the Prevention of Atrial Fibrillation After Cardiac Surgery: A Randomized Placebo-Controlled Trial
Brief Title: A Study of Stellate Ganglion Block for Prevention of Atrial Fibrillation
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erica D. Wittwer, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22-001106
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stellate ganglion block with local anesthetic (Experimental): Subjects will receive a single injection of bupivacaine in a stellate ganglion block
  Interventions: Procedure: Stellate ganglion block; Drug: Bupivacaine
- Stellate ganglion block with saline placebo (Sham Comparator): Subjects will receive a single injection of saline in a stellate ganglion block
  Interventions: Procedure: Stellate ganglion block; Drug: Placebo

INTERVENTIONS:
Procedure: Stellate ganglion block — Ultrasound guided injection into the stellate ganglion performed in the right side of the neck in a sterile fashion.
Drug: Bupivacaine — 10 mL of 0.5% without epinephrine injected in the plane of the right stellate ganglion
  Arms: Stellate ganglion block with local anesthetic
Drug: Placebo — 10 mL of saline injected in the plane of the right stellate ganglion
  Arms: Stellate ganglion block with saline placebo

SUMMARY:
The purpose of this study is to test if a nerve block procedure called a stellate ganglion block can help decrease the chance of atrial fibrillation after surgery. Atrial fibrillation is the abnormal, fast beating of the upper chambers of the heart. Stellate ganglion blockade has shown to decrease other types of abnormal heart rhythms as well as decrease the chance of atrial fibrillation.

DETAILED DESCRIPTION:
The investigator hypothesizes that stellate ganglion blockade with local anesthetic performed prior to cardiac surgery will reduce the incidence and duration of postoperative atrial fibrillation (POAF).

Specific Aim 1: Determine the incidence of POAF in patients receiving pre-surgical stellate ganglion blockade with local anesthetic versus saline placebo within one week of surgery or during hospitalization if discharged prior to one week.

Specific Aim 2: Determine the duration of POAF in patients receiving pre-surgical stellate ganglion blockade with local anesthetic versus saline placebo within one week of surgery or during hospitalization if discharged prior to one week.

Specific Aim 3: Determine the success rate of the block as evaluated by ipsilateral hand temperature change and skin sympathetic nerve activity (SKNA).

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting for cardiac surgery at the Mayo Clinic in Rochester, Minnesota.
* Patients scheduled to undergo mitral or aortic valve surgery with or without coronary artery bypass grafting.

Exclusion Criteria:

* Patients with a history of permanent atrial fibrillation, left or right ventricular assist device implantation or explantation.
* Patients with procedures not requiring cardiopulmonary bypass.
* Patients with procedures requiring deep hypothermic circulatory arrest.
* Patients with active infection or sepsis.
* Pre-operative immunosuppressive medication use (including steroid use).
* Pre-operative anti-arrhythmic medication use (aside from beta-blockers).
* Patients with Immunodeficiency syndrome.
* Patients with known neurologic disorder.
* Patients requiring left internal jugular central line placement.
* Performance of Maze procedures or left atrial appendage ligation procedures will not exclude patients from potential enrollment as atrial fibrillation still occurs postoperatively while the scarring from the Maze procedure forms.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of atrial fibrillation | Within one week of surgery or during hospitalization if discharged prior to one week
  Percentage of subjects to experience postoperative atrial fibrillation (POAF)

SECONDARY OUTCOMES:
Duration of atrial fibrillation | Within one week of surgery or during hospitalization if discharged prior to one week
  Duration of postoperative atrial fibrillation (POAF)
Skin Sympathetic Nerve Activity | 10-30 minute following performance of nerve block
  Measurement of difference in skin sympathetic nerve activity following block

CONTACTS AND LOCATIONS:
Overall Officials: Erica Wittwer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials